CLINICAL TRIAL: NCT04419246
Title: The Effect of Intravenous Tranexamic Acid and Interscalene Block Applied on Shoulder Arthroscopy on Total Blood Loss; a Prospective, Randomized, Controlled Trial
Brief Title: The Effect of Intravenous Tranexamic Acid and Interscalene Block Applied on Shoulder Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator ,Assoc. PhD. M.D., Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bursa BYIERH
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Nerve Block; Tranexamic Acid
MeSH Terms: interventions — Tranexamic Acid; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): interscalene block + General anesthesia
  Interventions: Other: interscalene block; Other: general anesthesia
- Group T (Active Comparator): Tranexamic acid +General anesthesia
  Interventions: Drug: tranexamic acid; Other: general anesthesia
- Group S (Sham Comparator): General anesthesia
  Interventions: Other: general anesthesia

INTERVENTIONS:
Other: interscalene block — ultrasound guided ultrasound guided interscalene block 30 minutes before operation. 30 minutes before operation.
  Arms: Group I
Drug: tranexamic acid — 10 mg/kg intravenous tranexamic acid 10 minutes before the incision.
  Arms: Group T
Other: general anesthesia — general anesthesia will be applied in accordance with standard procedures

SUMMARY:
Nerve blocks are used for pain and surgery after many operations today. It has been demonstrated by studies that the amount of postoperative bleeding decreases. On the other hand, surgical teams can use additional medications, such as Tranexamic acid, which have been proven by different studies that have reduced bleeding during and after arthroscopic surgery.

DETAILED DESCRIPTION:
The investigators aimed to investigate the effect of interscalene block application and tranexamic acid on bleeding in shoulder arthroscopy operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class
* underwent elective shoulder arthroscopy
* Patients with consent to participate in the study

Exclusion Criteria:

* history of arterial or venous thromboembolic disease
* Bleeding diathesis disorder
* Allergy to local anesthetics
* cardiac stent placement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2020-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
serum hemoglobin exchange | preoperative, postoperative 1st and 2nd day
  change of serum hemoglobin before and after operation

SECONDARY OUTCOMES:
postoperative bleeding amount | postoperative 24 hours
  The volume of drainage
Visual Analog Scale | Postoperative 24 hours
  Visual Analog Scale was used for pain.Pain intensity was measured using 0-10 cm visual analogue scale (VAS). (0= no pain, 10=intolerable pain)